CLINICAL TRIAL: NCT02713568
Title: Estimation of Fetal Weight by MR Imaging to PREdict Neonatal MACROsomia (PREMACRO Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Jani Jacques, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CHUB-PREMACRO
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Fetal Macrosomia
Keywords: Macrosomia; Magnetic Resonance- Estimated Fetal Weight; Ultrasound-Estimated Fetal Weight; Large-for-date fetus
MeSH Terms: conditions — Fetal Macrosomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Active Comparator): During routine third trimester ultrasound scan between 30 weeks and 35 weeks +6 days of gestational age, all women with an apparently normal, live singleton pregnancy, planning to deliver at the investigator's hospital maternity, will be invited to participate in the study.
  An Ultrasound scan to estimate the fetal weigth will be carried out during the 36th week of gestation.
  Interventions: Other: Ultrasound examination
- Magnetic Resonance (Experimental): During routine third trimester ultrasound scan between 30 weeks and 35 weeks +6 days of gestational age, all women with an apparently normal, live singleton pregnancy, planning to deliver at the investigator's hospital maternity, will be invited to participate in the study.
  A Magnetic Resonance examination to estimate the fetal weigth will be carried out during the 36th week of gestation.
  Interventions: Other: Magnetic resonance examination

INTERVENTIONS:
Other: Ultrasound examination — Prenatal Ultrasound examinations will be carried out using transabdominal sonography only by experienced consultants in MFM. Ultrasound-Estimated Fetal Weight will be obtained between 36.0-36.6 weeks of gestation, according to Hadlock et al.
  Operators performing the Ultrasound-Estimated Fetal Weight will be blinded to the results of Magnetic Resonance-Estimated Fetal Weight. The participants, general practitioners, obstetricians and midwifes of the patients will be aware of the results of Ultrasound-Estimated Fetal Weight which will be used for clinical management.
  For the primary outcome measure, macrosomia during Ultrasound-Estimated Fetal Weight will be defined as ≥ P95 based on Yudkin et al. For secondary outcome measures, it will be redefined as ≥ P90 or ≥ P99 based on Yudkin.
  Arms: Ultrasound
Other: Magnetic resonance examination — MRI will be performed the same day as the Ultrasound examination, using a clinical 1.5T whole-body unit.
  Operators performing Fetal Body Volume measurements will be blinded from Ultrasound-Estimated Fetal Weight results. Magnetic Resonance-Estimated Fetal Weight will be calculated using the equation 0,12+1,031*Fetal Body Volume = MR imaging weight (g) developed by Baker.
  General practitioners, obstetricians and midwifes of the patients will be blinded to the results of the Magnetic Resonance-Estimated Fetal Weight.
  For the primary outcome measure, macrosomia will be defined as ≥ P95 based on Yudkin et al. For secondary outcome measures, it will be defined as ≥ P90 or ≥ P99.
  Arms: Magnetic Resonance

SUMMARY:
Macrosomia and growth restriction are important causes of perinatal morbidity, at or near to term. However, clear identification of 'at risk' foetuses is difficult and clinical estimates of fetal weight are poor. Historically, ultrasound has been used as a second line in such cases but the accuracy of this imaging modality in the mid- to late third trimester is also limited.

Estimated fetal weight (EFW) is an important part of the clinical assessment and is used to guide obstetric interventions, when a fetus is small or large for dates. It frequently is the single most important component guiding interventions, such as induction of labour or Caesarean section.

Due to the imprecision of ultrasound-derived EFW, particularly in cases of suspected macrosomia in the 3rd trimester, the investigators believe that these estimates should not be used to make important obstetric decisions regarding mode and timing of delivery and that a more accurate method of assessment could produce better outcomes by restricting interventions to those foetuses at greatest risk. Some publications have already demonstrated that magnetic resonance (MR) imaging derived-EFW close to delivery, is more accurate than ultrasound

The goal of the present study is thus to compare the performance of magentic resonance imaging derived-EFW, versus ultrasound derived-EFW at 36 weeks of gestation, regarding the prediction of neonatal macrosomia.

DETAILED DESCRIPTION:
Macrosomia and growth restriction are important causes of perinatal morbidity, at or near to term. However, clear identification of 'at risk' foetuses is difficult and clinical estimates of fetal weight are poor. Historically, ultrasound has been used as a second line in such cases but the accuracy of this imaging modality in the mid- to late third trimester is also limited.

Estimated fetal weight (EFW) is an important part of the clinical assessment and is used to guide obstetric interventions, when a fetus is small or large for dates. When a diagnosis of intra-uterine growth restriction (IUGR) is made, the decision-making process is complex, particularly at very early gestations and involves multiple different factors, including maternal status, cardiotocography, liquor volume and dopplers. However, a large body of research is now available to assist with the management of both early and late-onset intrauterine growth restriction (IUGR) but there is a paucity of evidence to guide clinical practice, once macrosomia has been diagnosed, therefore the EFW is frequently the single most important component guiding interventions, such as induction of labour or Caesarean section.

Fetal macrosomia is associated with a higher incidence of perinatal morbidity, including shoulder dystocia and brachial plexus injury in the fetus and anal sphincter tears, uterine atony and haemorrhage in the mother. A recent multicentre randomised controlled trial appears to confirm the advantages of a policy of induction of labour for suspected macrosomia, demonstrating a clear reduction in the rates of shoulder dystocia and composite perinatal morbidity. However, some earlier but lower quality, observational studies have questioned the benefit of EFW made by ultrasonography in the last trimester, for suspected macrosomia, demonstrating that this practice can increase the risk of caesarean and instrumental delivery, without reducing perinatal morbidity.

Despite this conflicting data and a lack of evidence to support routine third trimester ultrasound, the absence of specific guidance, coupled with concerns regarding perinatal outcomes,mean that obstetricians will increasingly request an ultrasound at around 34-36 weeks gestation to identify foetuses above the 90th or below the 10th centiles. This practice will inevitably lead to increased and potentially harmful interventions based on relatively inaccurate data.

Due to the imprecision of ultrasound-derived EFW, particularly in cases of suspected macrosomia in the 3rd trimester, the investigators believe that these estimates should not be used to make important obstetric decisions regarding mode and timing of delivery and that a more accurate method of assessment could produce better outcomes by restricting interventions to those foetuses at greatest risk. Some publications have already demonstrated that magnetic resonance (MR) imaging derived-EFW close to delivery, is more accurate than ultrasound, with a mean percentage error superior to that of ultrasound and a recent meta-analyses has confirmed this promising accuracy.

The goal of the present study is thus to compare the performance of magentic resonance imaging derived-EFW, versus ultrasound derived-EFW at 36 weeks of gestation, regarding the prediction of neonatal macrosomia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects is ≥ 18 years of age and able to provide a written informed consent.
* Subject is a pregnant woman carrying a live singleton fetus at the 36+0-36+6 weeks scan, with no major abnormalities appearing during prenatal imaging with no major abnormalities appearing during prenatal imaging potentially affecting the correct use of the Hadlock formula for US-EFW. Conditions such as congenital diaphragmatic hernia with decreased abdominal circumference could be underestimated by the Hadlock USEFW. Another example is a massive sacro-coccygial teratomas.
* Subject is planning a delivery at our maternity at the University Hospital Brugmann, in Brussels, Belgium.
* Subject is known not to have any contra-indication to undergo an MR imaging examination.

Exclusion Criteria:

* Subject is known to have a contra-indication to undergo an MR imaging examination such as: Carrying a pacemaker or a metallic cardiac valve, having metallic material inside the head, having metallic fragments inside the eye following an accident, having any type of implant including ear implant, having a hip prosthesis
* Subject presenting with painful regular uterine contractions or history of ruptured membranes.
* Subjects who are unconscious, severely ill, mentally handicapped or under the age of 18 years.
* If birth occurs before MR and US evaluation.
* If patients delivers outside our local maternity unit.
* If the neonate's weigh is not measured within 6 hours after birth for any reason, including the need for emergency care immediately after delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2413 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Curve (AUROC) for prediction of macrosomia (≥ P95) | Between 36 weeks and 36 weeks + 6 days of gestation
  AUROC for prediction of macrosomia (≥ P95 for gestational age; normal ranges of Yudkin et al.) with MR (4 mm ST (slice thickness)/ 20 mm gap) versus US using the Hadlock equation.

SECONDARY OUTCOMES:
Area Under the Receiver Operating Curve (AUROC) for prediction of macrosomia (≥ P90) | Between 36 weeks and 36 weeks + 6 days of gestation
  AUROC for prediction of macrosomia (≥ P90 for gestational age) with magnetic resonnance (4 mm slice thickness/20 mm gap) versus ultrasound.
Area Under the Receiver Operating Curve (AUROC) for prediction of macrosomia (≥ P99) | Between 36 weeks and 36 weeks + 6 days of gestation
  AUROC for prediction of macrosomia (≥ P99 for gestational age) with Magnetic Resonance (4 mm slice thickness/ 20 mm gap) versus Ultrasound.
Area Under the Receiver Operating Curve (AUROC) for prediction of macrosomia (≥ P97) | Between 36 weeks and 36 weeks + 6 days of gestation
  AUROC for prediction of macrosomia (≥ P97 for gestational age) with Magnetic Resonance (4 mm slice thickness/ 20 mm gap) versus Ultrasound.
Area Under the Receiver Operating Curve (AUROC) for prediction of macrosomia (Abdominal Circumference) | Between 36 weeks and 36 weeks + 6 days of gestation
  AUROC for prediction of macrosomia with Abdominal Circumference ≥ P90 for gestational age. Measured in cm with Ultrasound
Area Under the Receiver Operating Curve (AUROC) for prediction of 'Small for gestational age' (SGA) | Between 36 weeks and 36 weeks + 6 days of gestation
  Measured with Magnetic Resonnace (4 mm slice thickness)/ 20 mm gap) versus ultrasound.
Comparative prediction rate for significant shoulder dystocia | Between 36 weeks and 36 weeks + 6 days of gestation
  Ability of Magnetic Resonnace-Estimated Fetal Weight (+/- pelvimetric measurements) vs. Ultrasound-Estimated Fetal Weigth in predicting significant shoulder dystocia. Significant shoulder dystocia is defined clinically as difficulty with delivery of the shoulders that was not resolved by the McRoberts' manoeuvre (flexion of the maternal thighs), usually combined with suprapubic pressure. Manoeuvres whose use suggested significant shoulder dystocia were those involving rotation of the fetus to displace the anterior shoulder impacted behind the maternal pubic bone (Woods, Rubin, or Jacquemier manoeuvres). The definition also included births with an interval of 60 s or more between delivery of the head and the body.
Comparative prediction rate for maternal morbidity | Between 36 weeks and 36 weeks + 6 days of gestation
  Ability of Magnetic Resonance-Estimated Fetal Weigth (+/- pelvimetric measurements) vs. Ultrasound-Estimated Fetal Weigth in predicting maternal morbidity, defined as caesarean section, operative vaginal delivery (vacuum or forceps), postpartum haemorrhage (1000 mL or more), blood transfusion, and anal sphincter tear.
Comparative prediction rate for neonatal morbidity | Between 36 weeks and 36 weeks + 6 days of gestation
  Ability of Magentic Resonance-Estimated Fetal Weigth (+/- pelvimetric measurements) vs. Ultrasound-Estimated Fetal Weigth in predicting neonatal morbidity, defined as arterial cord blood pH less than 7.10, Apgar score at 5 min less than 7, and admission to the neonatal intensive-care unit.
Comparative prediction rate for neonatal hyperbilirubinaemia | Between 36 weeks and 36 weeks + 6 days of gestation
  Ability of Magentic Resonance-Estimated Fetal Weigth (+/- pelvimetric measurements) vs. Ultrasound-Estimated Fetal Weigth in predicting neonatal hyperbilirubinaemia, defined as a maximum value exceeding 350 mmol/L of blood bilirubin.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Jani, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] King JR, Korst LM, Miller DA, Ouzounian JG. Increased composite maternal and neonatal morbidity associated with ultrasonographically suspected fetal macrosomia. J Matern Fetal Neonatal Med. 2012 Oct;25(10):1953-9. doi: 10.3109/14767058.2012.674990. Epub 2012 Apr 17. PMID 22439605
- [Background] DeVore GR. The importance of the cerebroplacental ratio in the evaluation of fetal well-being in SGA and AGA fetuses. Am J Obstet Gynecol. 2015 Jul;213(1):5-15. doi: 10.1016/j.ajog.2015.05.024. PMID 26113227
- [Background] McIntire DD, Bloom SL, Casey BM, Leveno KJ. Birth weight in relation to morbidity and mortality among newborn infants. N Engl J Med. 1999 Apr 22;340(16):1234-8. doi: 10.1056/NEJM199904223401603. PMID 10210706
- [Background] Seravalli V, Baschat AA. A uniform management approach to optimize outcome in fetal growth restriction. Obstet Gynecol Clin North Am. 2015 Jun;42(2):275-88. doi: 10.1016/j.ogc.2015.01.005. PMID 26002166
- [Background] Boulvain M, Senat MV, Perrotin F, Winer N, Beucher G, Subtil D, Bretelle F, Azria E, Hejaiej D, Vendittelli F, Capelle M, Langer B, Matis R, Connan L, Gillard P, Kirkpatrick C, Ceysens G, Faron G, Irion O, Rozenberg P; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Induction of labour versus expectant management for large-for-date fetuses: a randomised controlled trial. Lancet. 2015 Jun 27;385(9987):2600-5. doi: 10.1016/S0140-6736(14)61904-8. Epub 2015 Apr 8. PMID 25863654
- [Background] Bricker L, Neilson JP. Routine ultrasound in late pregnancy (after 24 weeks gestation). Cochrane Database Syst Rev. 2000;(2):CD001451. doi: 10.1002/14651858.CD001451. PMID 10796263
- [Background] Bricker L, Neilson JP, Dowswell T. Routine ultrasound in late pregnancy (after 24 weeks' gestation). Cochrane Database Syst Rev. 2008 Oct 8;(4):CD001451. doi: 10.1002/14651858.CD001451.pub3. PMID 18843617
- [Background] Rouse DJ, Owen J, Goldenberg RL, Cliver SP. The effectiveness and costs of elective cesarean delivery for fetal macrosomia diagnosed by ultrasound. JAMA. 1996 Nov 13;276(18):1480-6. PMID 8903259
- [Background] Gupta M, Hockley C, Quigley MA, Yeh P, Impey L. Antenatal and intrapartum prediction of shoulder dystocia. Eur J Obstet Gynecol Reprod Biol. 2010 Aug;151(2):134-9. doi: 10.1016/j.ejogrb.2010.03.025. Epub 2010 Apr 27. PMID 20427112
- [Background] Zaretsky MV, Reichel TF, McIntire DD, Twickler DM. Comparison of magnetic resonance imaging to ultrasound in the estimation of birth weight at term. Am J Obstet Gynecol. 2003 Oct;189(4):1017-20. doi: 10.1067/s0002-9378(03)00895-0. PMID 14586347
- [Background] Malin GL, Bugg GJ, Takwoingi Y, Thornton JG, Jones NW. Antenatal magnetic resonance imaging versus ultrasound for predicting neonatal macrosomia: a systematic review and meta-analysis. BJOG. 2016 Jan;123(1):77-88. doi: 10.1111/1471-0528.13517. Epub 2015 Jul 29. PMID 26224221
- [Background] Yudkin PL, Aboualfa M, Eyre JA, Redman CW, Wilkinson AR. New birthweight and head circumference centiles for gestational ages 24 to 42 weeks. Early Hum Dev. 1987 Jan;15(1):45-52. doi: 10.1016/0378-3782(87)90099-5. PMID 3816638
- [Background] Hadlock FP, Harrist RB, Carpenter RJ, Deter RL, Park SK. Sonographic estimation of fetal weight. The value of femur length in addition to head and abdomen measurements. Radiology. 1984 Feb;150(2):535-40. doi: 10.1148/radiology.150.2.6691115.
- [Background] Hadlock FP, Harrist RB, Sharman RS, Deter RL, Park SK. Estimation of fetal weight with the use of head, body, and femur measurements--a prospective study. Am J Obstet Gynecol. 1985 Feb 1;151(3):333-7. doi: 10.1016/0002-9378(85)90298-4. PMID 3881966
- [Background] Sampson ML, Gounden V, van Deventer HE, Remaley AT. CUSUM-Logistic Regression analysis for the rapid detection of errors in clinical laboratory test results. Clin Biochem. 2016 Feb;49(3):201-7. doi: 10.1016/j.clinbiochem.2015.10.019. Epub 2015 Oct 30. PMID 26523981
- [Background] Wani S, Hall M, Wang AY, DiMaio CJ, Muthusamy VR, Keswani RN, Brauer BC, Easler JJ, Yen RD, El Hajj I, Fukami N, Ghassemi KF, Gonzalez S, Hosford L, Hollander TG, Wilson R, Kushnir VM, Ahmad J, Murad F, Prabhu A, Watson RR, Strand DS, Amateau SK, Attwell A, Shah RJ, Early D, Edmundowicz SA, Mullady D. Variation in learning curves and competence for ERCP among advanced endoscopy trainees by using cumulative sum analysis. Gastrointest Endosc. 2016 Apr;83(4):711-9.e11. doi: 10.1016/j.gie.2015.10.022. Epub 2015 Oct 26. PMID 26515957
- [Background] Baker PN, Johnson IR, Gowland PA, Hykin J, Harvey PR, Freeman A, Adams V, Worthington BS, Mansfield P. Fetal weight estimation by echo-planar magnetic resonance imaging. Lancet. 1994 Mar 12;343(8898):644-5. doi: 10.1016/s0140-6736(94)92638-7. PMID 7906814
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- [Background] Leisenring W, Alonzo T, Pepe MS. Comparisons of predictive values of binary medical diagnostic tests for paired designs. Biometrics. 2000 Jun;56(2):345-51. doi: 10.1111/j.0006-341x.2000.00345.x. PMID 10877288
- [Derived] Kadji C, Cannie MM, Carlin A, Jani JC. Protocol for the prospective observational clinical study: estimation of fetal weight by MRI to PREdict neonatal MACROsomia (PREMACRO study) and small-for-gestational age neonates. BMJ Open. 2019 Mar 27;9(3):e027160. doi: 10.1136/bmjopen-2018-027160. PMID 30918039
- [Derived] Kadji C, Cannie MM, Resta S, Guez D, Abi-Khalil F, De Angelis R, Jani JC. Magnetic resonance imaging for prenatal estimation of birthweight in pregnancy: review of available data, techniques, and future perspectives. Am J Obstet Gynecol. 2019 May;220(5):428-439. doi: 10.1016/j.ajog.2018.12.031. Epub 2018 Dec 22. PMID 30582928